CLINICAL TRIAL: NCT02927314
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose-Finding Study of the Efficacy and Safety of CF102 in the Treatment of Non-Alcoholic Fatty Liver Disease (NAFLD) and Non-Alcoholic Steatohepatitis (NASH)
Brief Title: A Study of the Efficacy and Safety of CF102 in the Treatment of Non-Alcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Can-Fite BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CF102-211LD
Record Dates: First submitted 2016-09-25; First posted 2016-10-07 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Non-alcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — 2-chloro-N(6)-(3-iodobenzyl)adenosine-5'-N-methyluronamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo tablets orally q12h
  Interventions: Drug: Placebo
- CF102 12.5mg (Active Comparator): CF102 tablets orally q12h
  Interventions: Drug: CF102
- CF102 25mg (Active Comparator): CF102 tablets orally q12h
  Interventions: Drug: CF102

INTERVENTIONS:
Drug: CF102 — orally q12h
  Other Names: Cl-IB-MECA
  Arms: CF102 12.5mg; CF102 25mg
Drug: Placebo — orally q12h
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled clinical trial in subjects with NAFLD and NASH.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled study in subjects with a diagnosis of NAFLD. Subjects will undergo Screening procedures during the 4 weeks preceding Baseline. Subjects will be randomly assigned in a 1:1:1 ratio to oral doses of CF102 12.5 mg BID, CF102 25 mg BID, or matching placebo BID for 12 weeks using a stratified randomization, with stratification by presence or absence of diabetes mellitus. Subjects will be evaluated regularly for safety, and indicators of efficacy will be measured at Baseline and Week 12. Subjects will return for a follow-up visit 4 weeks after completion of the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Diagnosis of NAFLD by non-invasive determination of liver triglyceride concentration, as defined as triglyceride concentration ≥10.0% by NMRS.
3. At least 2 of the following:

   * Obesity, defined as body mass index (BMI) of ≥25 and ≤40 kg/m2; or waist circumference >88 and <200 cm for women or >102 and <200 cm for men
   * Type II diabetes mellitus, defined by the criteria of the American Diabetes Association (Appendix 1)
   * Blood pressure of 130/85 or higher (either systolic or diastolic)
   * Hypertriglyceridemia, defined as >150 mg/dL (>1.7 mmol/L)
   * Reduced high-density lipoprotein (HDL) cholesterol, defined as <40 mg/dL (<1.04 mmol/L) in men or <50 mg/dL (<1.3 mmol/L) in women.
4. Acceptable hepatic metabolic and synthetic function, as indicated at Screening by:

   * Serum albumin ≥3.5 gm/dL
   * INR ≤1.2
   * Serum total bilirubin ≤2.0 mg/dL.
5. Absence of cirrhosis, defined as a Fibroscan score of ≤F4 and liver stiffness measurement (LSM) of 7 13 kPa.
6. The following laboratory values must be documented at Screening prior to initiation of study drug:

   * Absolute neutrophil count >1.5x109/L
   * Platelet count >100x109/L
   * Serum creatinine <2.0 mg/dL.
7. For women of childbearing potential, negative serum pregnancy test result (not pregnant or lactating).
8. Understand and provide written informed consent to participate.
9. Patients taking herbal supplements, homeopathic medications, or other alternative treatments, must be on a stable regimen for at least 6 months prior to randomization.
10. Willing to comply with scheduled visits, treatment plans, laboratory assessments, and other study-related procedures.

Exclusion Criteria:

1. Presence of ascites, hepatic encephalopathy, or other clinical evidence of cirrhosis.
2. Other active acute or chronic liver disease, such as autoimmune hepatitis, hepatitis B, hepatitis C, alcoholic liver disease, or hepatocellular carcinoma at the time of Screening and randomization.
3. Familial dyslipidemia.
4. Weight loss of >5% within 6 months prior to Baseline.
5. History of bariatric surgery within 5 years of Screening.
6. Diabetes mellitus other than Type II.
7. Daily alcohol intake >20 g/day for women and 30 g/day for men (on average per day), as per medical history.
8. Treatment with the following anti-diabetic medications: DPP-4 inhibitor unless it was stopped 3 months before Screening, GLP-1 receptor agonists (such as Januvia [sitagliptin], Byetta [incretin], etc.) unless it was started at least 12 months and on stable dose at least 3 months prior to Screening.
9. Metformin, fibrates, statins, insulin, or sulfonylurea unless the dose has been stabilized for the last 1 month prior to Screening.
10. More than 7 days of treatment with valproic acid, tamoxifen, methotrexate, amiodarone, rifaximin, other antibiotics, or anti-cholinergic agents within 3 months prior to Screening.
11. Uncontrolled or clinically unstable thyroid disease, in the judgment of the Principal Investigator.
12. Seropositivity for markers of viral hepatitis or human immunodeficiency virus (HIV) at Screening.
13. Uncontrolled arterial hypertension or congestive heart failure (New York Heart Association Classification 3 or 4).
14. Angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism within 3 months prior to initiation of study drug.
15. History of or ongoing cardiac dysrhythmias requiring treatment, atrial fibrillation of any grade, or persistent prolongation of the QTc (Fridericia) interval to >450 msec for males or >470 msec for females.
16. Pregnant or lactating female.
17. Women of childbearing potential, unless they agree to use dual contraceptive methods which, in the opinion of the Principal Investigator, are effective and adequate for that patient's circumstances while on study drug.
18. Men who partner with a woman of childbearing potential, unless they agree to use effective, dual contraceptive methods (ie, a condom, with female partner using oral, injectable, or barrier method) while on study drug.
19. Any severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, may interfere with the informed consent process and/or with compliance with the requirements of the study, or may interfere with the interpretation of study results and, in the investigator's opinion, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of CF102 as determined by change in serum alanine aminotransferase (ALT) levels | 12 weeks
  Mean percent change in serum alanine aminotransferase (ALT) levels
Efficacy of CF102 as determined by change in magnetic resonance imaging-determined hepatic steatosis | 12 weeks
  Percent change from Baseline in hepatic steatosis measured by magnetic resonance imaging-determined proton-density fat-fraction (MRI-PDFF)

SECONDARY OUTCOMES:
Body weight in subjects with NAFLD | 12 weeks
  Change from baseline in body weight (kg)
Waist circumference in subjects with NAFLD | 12 weeks
  Change from baseline in waist circumference (cm)
HDL cholesterol levels in subjects with NAFLD | 12 weeks
  Change from baseline in serum triglyceride and HDL cholesterol levels (mg/dL)
Normalization of serum ALT levels in subjects with NAFLD | 12 weeks
  Proportion of all subjects whose serum ALT level normalizes
Serum aspartate aminotransaminase (AST) levels in subjects with NAFLD | 12 weeks
  Change from baseline in serum AST levels
Hemoglobin A1c levels and degree of insulin resistance | 12 weeks
  Change from baseline in Homeostasis Model Assessment (HOMA)
Pharmacokinetics (PK) of CF102 in this population | 12 weeks
  PK of CF102 will be assessed through steady state trough drug level
Peripheral blood expression of the A3 adenosine receptor (A3AR). | 12 weeks
  Change from baseline in A3 adenosine receptor (A3AR) expression level
Nature, frequency, and severity of adverse events in this patient population | 12 weeks
  Nature, frequency, and severity (by CTCAE or comparable scale) of adverse events

OTHER OUTCOMES:
Serum adiponectin levels | 12 weeks
  Change from baseline in serum adiponectin levels in subjects with NAFLD
Serum leptin levels | 12 weeks
  Change from baseline in serum leptin levels in subjects with NAFLD
Serum alpha-2 macroglobulin levels | 12 weeks
  Change from baseline in serum alpha-2 macroglobulin levels in subjects with NAFLD
Serum apolipoprotein A1 levels | 12 weeks
  Change from baseline in serum apolipoprotein A1 levels in subjects with NAFLD
Serum haptoglobin levels | 12 weeks
  Change from baseline in serum haptoglobin levels in subjects with NAFLD
Serum C-reactive protein levels | 12 weeks
  Change from baseline in serum C-reactive protein levels in subjects with NAFLD
Liver stiffness | 12 weeks
  Change from baseline in liver stiffness by FibroScan in subjects with NAFLD

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Silverman, MD, Study Director — Can-Fite BioPharma Ltd
Locations (3):
- Israel (3):
  - Can-Fite Investigational Site #318, Jerusalem
  - Can-Fite Investigational Site #319, Nazareth
  - Can-Fite Investigational Site #311, Petah Tikva

REFERENCES:
- [Derived] Muthiah MD, Siddiqui MS. Editorial: targeting aberrant hepatic inflammation for treatment of non-alcoholic steatohepatitis. Aliment Pharmacol Ther. 2022 Feb;55(4):483-484. doi: 10.1111/apt.16748. No abstract available. PMID 35092056
- [Derived] Safadi R, Braun M, Francis A, Milgrom Y, Massarwa M, Hakimian D, Hazou W, Issachar A, Harpaz Z, Farbstein M, Itzhak I, Lev-Cohain N, Bareket-Samish A, Silverman MH, Fishman P. Randomised clinical trial: A phase 2 double-blind study of namodenoson in non-alcoholic fatty liver disease and steatohepatitis. Aliment Pharmacol Ther. 2021 Dec;54(11-12):1405-1415. doi: 10.1111/apt.16664. Epub 2021 Oct 20. PMID 34671996